CLINICAL TRIAL: NCT02624141
Title: Open Multicentric Study to Assess the Hematopoyetic Response in Terms of Increase of Hemoglobin Levels, of Patients With Anemia Reklated to Malignant Tumors, Treated With Erythropoietin B (Recormon) Using the Pre-Filled Syringe With 30,000 IU, as Well as to Quantify Teh Risk Factors of Anemia and Its Impact on Quality of Life Related to Treatment
Brief Title: A Study of Recormon (Epoetin Beta) in Anemic Patients With Non-Myeloid Malignancy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to low recruitment
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18054
Record Dates: First submitted 2015-12-02; First posted 2015-12-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

ARMS (1):
- Epoetin Beta 30000 IU (Experimental): Dosage at Initiation: Subcutaneous injection of 30000 IU epoetin beta administered once a week. Dosage could be increased to 30000 IU twice a week or 60000 IU once a week after 4 weeks.
  Interventions: Drug: Epoetin Beta

INTERVENTIONS:
Drug: Epoetin Beta — Dosage at Initiation: Subcutaneous injection of 30000 IU administered once a week. Dosage could be increased to 30000 IU twice a week or 60000 IU once a week after 4 weeks if a blood transfusion was required or hemoglobin level did not increase by at least 0.5 grams per deciliter (g/dL) versus baseline.
  Other Names: Recormon

SUMMARY:
This study will examine the efficacy, safety, and effect on hemoglobin levels, of once weekly epoetin beta subcutaneous injections (30,000 International Units [IU]) in anemic patients with solid tumors. The anticipated study duration is 4 months, and the target sample size is 40 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a non-myeloid malignancy
* Anemia

Exclusion Criteria:

* Transfusion of red blood cells within 2 months of study drug
* Treatment-resistant hypertension
* Acute or chronic bleeding (requiring therapy) within 3 months of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin Levels at 16 Weeks | 16 Weeks

SECONDARY OUTCOMES:
Serum Iron Levels | 16 Weeks
Quality of Life According to Functional Assessment of Cancer Therapy - Anemia (FACT-An) Instrument | Up to 4 months
Tolerability - Incidence of Adverse Events | Up to 4 months
Serum Transferrin Levels | 16 Weeks
Percentage of Participants With A Positive Response | 16 Weeks
Time To Global Response | Up to 4 months
Quality of Life In Relation to Anemia Grade | Up to 4 months
Serum Ferritin Levels | 16 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (2):
- Venezuela (2):
  - Caracas
  - Valencia